CLINICAL TRIAL: NCT01668251
Title: National Collaborative Study of Girls Prenatally Diagnosed With Turner Syndrome Karyotypes
Brief Title: Turner Syndrome Prenatal Diagnosis Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Patricia Fechner, Associate Professor, Pediatrics, Seattle Children's Hospital
Other Study IDs: TS Prenatal Study
Record Dates: First submitted 2011-11-03; First posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Turner Syndrome
Keywords: Turner syndrome; Diagnosis, prenatal
MeSH Terms: conditions — Turner Syndrome; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fetal ascertainment: Girls who are diagnosed with Turner syndrome because of concerns raised by an abnormal fetal ultrasound.
- Maternal ascertainment: Girls who are diagnosed with Turner syndrome because their mothers had an amniocentesis for a reason other than an abnormal fetal ultrasound concerning for Turner syndrome. For example an amniocentesis was done because of advanced maternal age or because of an abnormal triple screen or because another condition was being screened for such as trisomy 21.

SUMMARY:
The goal of this study is to compare the features of Turner syndrome in girls who are diagnosed before birth because of fetal concerns versus those who are diagnosed when their mother has an amniocentesis for another reason.

DETAILED DESCRIPTION:
This is an observational study which will look at girls who are diagnosed with Turner syndrome before they are born. Girls will be divided into two groups: 1) those diagnosed because of features seen on ultrasound which raised the question of Turner syndrome and 2) those diagnosed incidentally when their mother had an amniocentesis for another reason such as advanced maternal age.

No clinical procedures nor interventions will be done as part of this data collection study which will occur for the first 3 to 6 years of the girl's life. The investigators will be looking to see if girls who are diagnosed incidentally have less features of Turner syndrome than those girls who are diagnosed because of fetal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Turner syndrome diagnosed prenatally
* Less than 4 months of age at time of enrollment

Exclusion Criteria:

* Turner syndrome diagnosed postnatally
* Older than 4 months of age at time of enrollment

Max Age: 3 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: Girls who are diagnosed with Turner syndrome prenatally.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2006-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Number of signs of Turner syndrome | three to six years
  Girls diagnosed with Turner syndrome by fetal ascertainment will have more signs of Turner syndrome than girls diagnosed by maternal ascertainment

SECONDARY OUTCOMES:
Growth | three to six years
  Do girls with Turner syndrome ascertained by fetal ascertainment grow differently than girls ascertained by maternal ascertainment.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Fechner, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Background] Gunther DF, Eugster E, Zagar AJ, Bryant CG, Davenport ML, Quigley CA. Ascertainment bias in Turner syndrome: new insights from girls who were diagnosed incidentally in prenatal life. Pediatrics. 2004 Sep;114(3):640-4. doi: 10.1542/peds.2003-1122-L. PMID 15342833